CLINICAL TRIAL: NCT05089461
Title: An Open-label, Multi-center Phase II Clinical Trial to Evaluate the Cardiac Safety of Mitoxantrone Hydrochloride Liposome Injection in the Treatment of Advanced Malignant Tumor
Brief Title: A Study to Evaluate the Cardiac Safety of Mitoxantrone Hydrochloride Liposome Injection in the Treatment of Advanced Malignant Tumor
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decided to stop
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-020
Record Dates: First submitted 2021-10-09; First posted 2021-10-22 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): Patients with advanced malignant tumor will receive 20 mg/m^2 Mitoxantrone Hydrochloride Liposome by an intravenous infusion (IV) on day 1 of each treatment cycle.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome — Mitoxantrone Hydrochloride Liposome, intravenous injection (IV), 20 mg/m^2. Solid tumors: every 3 weeks (q3w, 1 cycle), Lymphoma: every 4 weeks (q4w, 1 cycle).

SUMMARY:
This is a multicenter, open-label, phase II study to evaluate the cardiac safety of Mitoxantrone Hydrochloride Liposome in patients with advanced malignant tumor who has received at least first-line treatment.

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase II study to evaluate the cardiac safety of Mitoxantrone Hydrochloride Liposome in patients with advanced malignant tumor who has received at least first-line treatment. About 120 patients will be recruited in this study. Patients with solid tumors will receive Mitoxantrone Hydrochloride Liposome 20 mg/m^2 by an intravenous infusion (IV) every 3 weeks (q3w, 1 cycle). Patients with lymphoma will receive Mitoxantrone Hydrochloride Liposome 20 mg/m^2 by an intravenous infusion (IV) every 4 weeks (q4w, 1 cycle). All the patients will receive the treatment until disease progression, intolerable toxic reaction, death, or withdrawal by investigator's or patient's decision.

ELIGIBILITY:
Inclusion Criteria:

1. Patients fully understand and voluntarily participate in this study and sign informed consent;
2. Age ≥18 years;
3. Histologically confirmed diagnosis of late-stage solid tumor or peripheral T cell lymphoma (PTCL);
4. Has received standard first-line treatment;
5. Previous treated with anthracyclines, and converted to doxorubicin at equivalent doses. The cumulative dose of doxorubicin is 160 mg/m^2 < doxorubicin ≤550 mg/m^2;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
7. Adequate organ function:

   * Absolute neutrophil count (ANC) >1.5 10^9/L;
   * Hemoglobin > 90 g/L;
   * Platelet count > 75 10^9/L;
   * Creatinine < 1.5 upper limit of normal (ULN);
   * Total bilirubin < 1.5 ULN (< 3 ULN in patients with hepatic metastasis);
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 ULN (< 5 ULN in patients with hepatic metastasis);
8. Patients of childbearing potential must agree to use effective contraceptive measures from screening until 6 months after the end of the last dose; Female patients must have a negative pregnancy test before enrolment.

Exclusion Criteria:

1. History of allergy to mitoxantrone hydrochloride or liposomal drugs;
2. Other malignant tumors in the past 3 years, excluding cervical carcinoma in situ, basal cell carcinoma of the skin or squamous cell carcinoma of the skin that have been radically treated;
3. Cerebral or meningeal metastases;
4. HBsAg or HBcAb positive with HBV DNA ≥ 2000 IU/mL, HCV antibody positive with HCV RNA above the lower limit of detection of the study center, or human immunodeficiency virus (HIV) antibody positive;
5. Life expectancy ≤ 12 weeks;
6. AEs from the previous treatment > Grade 1 based on CTCAE (except for the toxicity without safety risk judged by the investigator, such as alopecia, hyperpigmentation);
7. Cardiac dysfunction, including:

1)Long QT interval syndrome; 2)High-degree atrioventricular block; 3)Malignant arrhythmia poorly controlled by medication; 4)A history of chronic heart failure with NYHA≥3; 5)Severe heart valve regurgitation or stenosis requiring treatment; 6)Acute coronary syndrome, severe pericardial disease, severe myocardial disease within 6 months prior to screening; 7)Poorly controlled hypertension (defined as systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than100 mmHg, measured ≥3 times, under control of antihypertensive drug); 8)Echocardiography showed LVEF < 50%; 8.Active bacterial or fungal infection requiring systemic intravenous therapy within 1 week before the first dose; 9.Use of other anticancer treatment within 4 weeks prior to the first dose; 10.Enrolled in any other clinical trials within 4 weeks prior to the first dose; 11.Patients underwent major surgery within 3 months prior to the first dose, or have a surgical schedule during the study period;; 12.Thrombosis or thromboembolism within 6 months prior to the first dose; 13.Lactating female; 14.Serious and/or uncontrolled systemic diseases; 15.Not suitable for this study as decided by the investigator due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac adverse event | up to approximately 5 years.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to approximately 3 years
Progression-free survival (PFS) | up to approximately 3 years.
Overall survival (OS) | up to approximately 5 years
Incidence of treatment emergent adverse event (TEAE) | up to approximately 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Dalian medical university, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No